CLINICAL TRIAL: NCT07094360
Title: Effect of Hydrotherapy on Performance in Children With Brain Tumor
Brief Title: Effect of Hydrotherapy on Children With Brain Tumor
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mahmoud Usama Mahmoud Ahmed, Lecturer at Pediatric department, Faculty of Physical Therapy, Cairo University., Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2490-2016
Record Dates: First submitted 2025-07-21; First posted 2025-07-30 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Pediatric Brain Tumor
Keywords: Hydrotherapy; Performance; Children; Brain tumor
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Land-based exercise program (Experimental): Land-based exercise program
  Interventions: Other: Land-based exercise program
- Hydrotherapy besides Land-based exercise program (Experimental): Hydrotherapy besides Land-based exercise program
  Interventions: Other: Hydrotherapy besides Land-based exercise program

INTERVENTIONS:
Other: Land-based exercise program — Land-based exercise program
  Arms: Land-based exercise program
Other: Hydrotherapy besides Land-based exercise program — Hydrotherapy besides Land-based exercise program
  Arms: Hydrotherapy besides Land-based exercise program

SUMMARY:
* Background: Brain and spinal cord tumors are the second most common cancers in children (after leukemia). They account for about 1 out of 4 childhood cancers. More than 4,000 central nervous system tumors are diagnosed each year in children and teens. (Blaney et al., 2011).
* Aim: It has been reported that those children have easy fatigability so the purpose of this study is to investigate the effectiveness of hydrotherapy on endurance in these Children.
* Significance: The effects of physical exercise training interventions for childhood cancer participants are not yet convincing due to small numbers of participants and insufficient study methodology. More and high-quality evidence is needed in order to be able to draft exercise and physical activity guidelines for this population. Despite the positive results of exercise interventions in adult cancer patients, the evidence for benefits in childhood cancer patients is limited (Braam et al., 2013).

An 8-week deep water exercise program was clinically effective for improving CRF(Cancer-Related-Fatigue), muscle strength, and several aspects of mood state as compared with usual treatment care at short and medium term in breast cancer survivors reporting a moderate rate of fatigue (Irene et al., 2013).

In this study, the investigators are trying to find out the effect of hydrotherapy as a way of fun and amusement that children can do easily with great pleasure and also as a treatment method.

* Subjects: Thirty children of both sexes will participate in this study. Inclusion criteria: Children between 5-14 years old after brain tumor resection surgery 2 weeks post-surgery. Exclusion Criteria: Cognitive or mental (developmental), or both, impairment, Children with a genetic disorder, Children with a chronic lung disease, Severe cardiomyopathy (ejection fraction <40%, ischemia and angina pectoris at rest), Children with a neuromuscular disease.
* Methodology:

For Evaluation: Lafayette manual muscle tester to assess muscle endurance/strength (Lafayette instrument evaluation, 2015). The pediatric quality of life inventory version 4(PedsQL) is used to assess quality of life (Varni et al., 1999). The nine-minute run-walk test (Guedes et al., 2006) and the timed up-and-down stairs test (Zaino et al., 2004) are to measure Cardiorespiratory fitness.

For Treatment: Children will be divided into two groups, control group will receive a land-exercise program and study group will receive the same exercise program then repetition of these exercises under water to study the effectiveness of using hydrotherapy. The program will take 30 minutes (5 minutes each with 1 minute rest in between).

The selected program will be in the form of:

1. Sitting while strengthening shoulder horizontal adductors by using weights.
2. Sitting while pushing down by using weights.
3. Sitting while strengthening elbow extensors by using weights.
4. Sitting while holding weights for a while.
5. Standing on uneven surface.
6. Pushing downs by legs.
7. Sitting balance.
8. Sitting with pushing by hands while making legs as glue.
9. Sitting with kicking by legs while fixing hands.
10. Standing and throwing a ball.
11. Weight shifting and recovery while initiating single limb support.

ELIGIBILITY:
Inclusion Criteria:

They will be selected according to the following criteria:

1. Children between 5-14 years old.
2. Children after brain tumor resection surgery 4 weeks post-surgery.

Exclusion Criteria:

Children who have one or more of the following criteria will be excluded from the study:

1. Children who cannot follow orders or instructions.
2. Children with a genetic disorder.
3. Children with a chronic lung disease.
4. Sever cardiomyopathy (ejection fraction <40%, ischemia and angina pectoris at rest).
5. Children with a neuromuscular disease.

Ages: 5 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Muscle strength of upper and lower limb muscles | 4-6 months
  Lafayette Manual Muscle Tester:
  The test was performed by applying force to the limb of a child as he/she resists the force isometrically. The objective of the test is for the clinician to overcome or "break" the child's resistance. When the resistance "break" occurs the Lafayette Manual Muscle Tester (MMT) records the peak force and the time required to achieve the "break providing reliable, accurate, and stable muscle strength readings that conform to most manual muscle testing protocols. The MMT also features a wide range of customizable options for data storage, preset test times, and force thresholds

SECONDARY OUTCOMES:
Pediatric quality of life | 4-6 months
  The pediatric quality of life inventory version 4 (PedsQL) is a modular approach to measure health-related quality of life in healthy children and adolescents and those with acute and chronic health conditions. The Pads Measurement Model integrates seamlessly both generic core scales and disease-specific modules into one measurement system. The PedsQL Brain tumor module was used in this study.
Cardiorespiratory fitness | 4-6 months
  The Six-minute run-walk test:
  This test has been used as an adaptation of the 12-minute Cooper test for children under the age of 12, and is also used in Brazil and internationally as an alternative to motor test batteries for CRF assessment (Gaya et al., 2007). Currently, it becomes modified to the 6-minute walk